CLINICAL TRIAL: NCT02337049
Title: Preeclampsia Subtypes and Surrogate Markers of CVD Risk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Randers Regional Hospital (Other); Karen Elise Jensen Foundation (Other); Central Denmark Region (Other)
Responsible Party: Sponsor
Other Study IDs: 26702017
Record Dates: First submitted 2015-01-05; First posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Preeclampsia
Keywords: Preeclampsia. Cardiovascular Disease (CVD) Risk.
MeSH Terms: conditions — Pre-Eclampsia; Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood serum. Blood plasma. Urine.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Previously early onset preeclampsia: Women with a history of early onset preeclampsia 10 years ago
- Previously late onset preeclampsia: Women with a history of late onset preeclampsia 10 years ago
- Previously normotensive pregnancy: Women with a history of normotensive pregnancies 10 years ago

SUMMARY:
In order to assess surrogate markers of cardiovascular risk in subtypes of preeclampsia, we will conduct a 10-year follow-up study comparing 40 women with a history of early onset preeclampsia; 40 women with a history of late onset preeclampsia and 40 women with a history of normotensive pregnancies.

Eligible participants delivered at the Department of Obstetrics at Randers Regional Hospital 1998-2008.

Early-onset preeclampsia is defined as preeclampsia that develops before 34 weeks of gestation, whereas late-onset preeclampsia develops at or after 34 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

* Women who delievered at the Department of Obstetrics at Randers Regional Hospital 1998-2008

Exclusion Criteria:

* Current pregnancy or breastfeeding

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible participants delivered at the Department of Obstetrics at Randers Regional Hospital 1998-2008. Early-onset preeclampsia is defined as preeclampsia that develops before 34 weeks of gestation, whereas late-onset preeclampsia develops at or after 34 weeks of gestation.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Echocardiographic Markers of Cardiac Strain | 10 years postpartum

SECONDARY OUTCOMES:
Markers of arteriosclerosis and atherosclerosis | 10 years postpartum
Circulating biomarkers of cardiovascular disease. | 10 years postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Ulla B Knudsen, Professor, Study Chair — Department of Obstetrics and Gynaecology, Aarhus University Hos; Martin Christensen, MD, Principal Investigator — Clinical Research Unit, Randers Regional Hospital; Camilla S Kronborg, MD, PhD, Study Director — Department of Oncology, Aarhus University Hospital
Locations (1):
- Randers Regional Hospital, Randers, Randers NØ, Denmark